CLINICAL TRIAL: NCT04286230
Title: Construct Validation of the BIOTICA Questionnaire (Barriers to Optimal Medication Adherence With Oral Antibiotics)
Brief Title: Construct Validation of the BIOTICA Questionnaire
Acronym: BIOTICA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00069
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Infectious Diseases and Manifestations
Keywords: Adherence; Oral antibiotics; Electronic monitoring
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Adherence to oral antibiotics assessed by Questionnaire — The purpose of the BIOTICA-questionnaire is to detect individual barriers preventing the optimal intake of oral antibiotics and thus, leading to inadequate adherence or persistence to the regimen.
Behavioral: Persistence to oral antibiotics assessed by Questionnaire — The purpose of the BIOTICA-questionnaire is to detect individual barriers preventing the optimal intake of oral antibiotics and thus, leading to inadequate adherence or persistence to the regimen.

SUMMARY:
Based on barriers identified in a systematic literature search, a self-report questionnaire called "BIOTICA" has been developed by the research team to assess medication adherence barriers to oral AB. The purpose of the BIOTICA-questionnaire is to detect individual barriers that prevent the optimal intake of oral AB and thus, lead to inadequate adherence or persistence to the regimen. A study is now needed to establish construct validity. Correlation between the answers to the BIOTICA-questionnaire and the electronically monitored intake of the oral AB will be analyzed in the general population.

DETAILED DESCRIPTION:
Global consumption of oral antibiotics (AB) is increasing, with 80% of all prescriptions in Europe stemming from primary care, mostly against respiratory tract infections. Adequate intake behavior (i.e. adherence) to oral AB is vital to prevent therapeutic failure, to reduce the risk of microbial resistance, to reduce health care consumption, medication waste and environmental pollution. However, non-adherence among oral AB users reaches rates of 21%-38% during an AB treatment course. To improve medication adherence, understanding patient barriers to treatment is crucial. Based on barriers identified in a systematic literature search, a self-report questionnaire called "BIOTICA" has been developed by the research team to assess medication adherence barriers to oral AB. The purpose of the BIOTICA-questionnaire is to detect individual barriers that prevent the optimal intake of oral AB and thus, lead to inadequate adherence or persistence to the regimen. A study is now needed to establish construct validity (also called criterion, convergent or concurrent validity) that is, to generate evidence that the questionnaire measures what it is intended to. Thus, the instrument under investigation (i.e. BIOTICA-questionnaire) will be distributed at the same time as the targeted attribute (i.e. adherence to oral AB) will be electronically monitored in the general population. The correlation between the two measurements will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* is ≥ 18 years
* has a prescription for an oral AB for 3-30 days
* self-manages medication
* is able to read and understand the German language
* signs the Informed Consent Form (ICF)
* accepts to record the intake of oral AB with the electronic device Time4Med™

Exclusion Criteria:

* is cognitively impaired
* is currently pregnant or actively trying to get pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The general population entering a community pharmacy.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence [%] to oral antibiotics | maximum 30 days
  The primary endpoint is the adherence [%] to oral antibiotics calculated as correct dosing days from the electronic adherence data

SECONDARY OUTCOMES:
Persistence [%] to oral antibiotics | maximum 30 days
  The secondary endpoint is persistence [%] to oral antibiotics defined as the time until medication discontinuation and calculated as the percentage of days with at least one intake

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arnet, Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Apotheke am Spalenbärg, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
csv files containing the de-identified patient adherence raw data will be forwarded on request
Time Frame: mid 2022
Access Criteria: on request to the principal investigator